CLINICAL TRIAL: NCT02722967
Title: A Multicenter, 8-week, Open-label, Single-Arm Exploratory Trial to Assess the Functionality of an Integrated Call Center for the Digital Medicine System by Adult Subjects With Schizophrenia, Major Depressive Disorder, or Bipolar 1 Treated With Oral Aripiprazole
Brief Title: Exploratory Trial to Assess the Functionality of an Integrated Call Center for the Digital Medicine System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316-13-215
Record Dates: First submitted 2016-03-13; First posted 2016-03-30 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bipolar I Disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole + IEM (Experimental): Subjects will receive an intervention consisting of a drug-device combination that consists of an aripiprazole tablet with a tiny sensor embedded within it referred to as an Ingestible Event Marker (IEM) . They will discontinue their normally prescribed oral aripiprazole tablets and will take the aripiprazole(2, 5, 10, 15, 20, or 30 mg) + IEM once daily for the 8-week assessment period for this trial.
  Interventions: Drug: Aripiprazole + IEM (Ingestible Event Marker)

INTERVENTIONS:
Drug: Aripiprazole + IEM (Ingestible Event Marker) — Oral aripiprazole (2, 5, 10, 15, 20, or 30 mg) with an ingestible event marker in a single daily dose for duration of the trial.
  Other Names: MIND1; Digital Medicine System

SUMMARY:
This study will assess the helpfulness of the integrated call center in optimizing use of the Digital Medicine System in adult subjects with Schizophrenia, Major Depressive Disorder, or Bipolar Disorder taking oral aripiprazole.

DETAILED DESCRIPTION:
The Digital Medicine System includes a drug-device combination of aripiprazole + an ingestible event marker (IEM), a wearable sensor (skin patch), and application software to convey the level of activity and rest, and to mark events through the act of ingestion.

Physician and self-report are the most commonly used to assess medication compliance yet studies have consistently found that healthcare providers' subjective judgments of medication compliance are often inaccurate, with a tendency for practitioners to overestimate subject adherence. The sponsor's intent is to develop a system that will benefit future subjects by providing the ability to measure their medication-taking behavior in an objective manner and being able to monitor several physiologic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Schizophrenia (SCH), Major Depressive Disorder (MDD), or Bipolar 1 Disorder (BP1), per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Must be able to swallow tablets
* Currently taking a stable daily dose of oral aripiprazole
* Must have capacity to utilize the technology
* Skin in area of patch application must be free of any skin disorders or dermatological problems

Exclusion Criteria:

* Subjects using long acting injectable antipsychotic medications
* Subjects likely to be incapable of using the Digital Medicine System even with assistance
* Subjects who present serious risk of suicide
* History of epilepsy or seizures
* History of hypersensitivity to antipsychotic agents, adhesive tape or any component of the sensor skin patch or ingestible event marker
* Current history of substance use disorder meeting DSM-5 criteria
* Subject with unstable mood, acute psychosis or exhibiting symptoms requiring hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Peters-Strickland, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (4):
- United States (4):
  - Granada Hills, California
  - Rochester, New York
  - Durham, North Carolina
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jan M, Coppin-Renz A, West R, Gallo CL, Cochran JM, Heumen EV, Fahmy M, Reuteman-Fowler JC. Safety Evaluation in Iterative Development of Wearable Patches for Aripiprazole Tablets With Sensor: Pooled Analysis of Clinical Trials. JMIR Form Res. 2023 Dec 12;7:e44768. doi: 10.2196/44768. PMID 38085556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, single-arm trial assessed the functionality of an integrated call center for digital medicine system (DMS) as used by adult subjects (18 to 65 years of age, inclusive, at the time of screening) with Schizophrenia (SCH), Bipolar 1 disorder (BP1), or Major depressive disorder (MDD) being treated with oral aripiprazole.
Pre-assignment Details: The trial consisted of a screening period of ≤ 7 days. This period assessed the eligibility criteria at 1 or more visits. An interactive web response system (IWRS) was used to obtain an identification number for each subject with a signed electronic informed consent form (eICF).
Groups:
- Bipolar 1 Disorder (BP1): This group consisted of the participants with acute treatment of manic and mixed episodes associated with BP1 who were being treated with oral aripiprazole.
- Major Depressive Disorder (MDD): This group consisted of the participants with adjunctive treatment of MDD who were being treated with oral aripiprazole.
- Schizophrenia (SCH): This group consisted of the participants with SCH who were being treated with oral aripiprazole.
Period: Overall Study
Arm/Group | Bipolar 1 Disorder (BP1) | Major Depressive Disorder (MDD) | Schizophrenia (SCH)
Started | 22 | 12 | 15
Completed | 17 | 10 | 11
Not Completed | 5 | 2 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Non-compliance with patch wearing | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Non-adherence of the patch to the skin | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Sample: All subjects who entered the trial and used Digital Medicine System (DMS).
Groups:
- Bipolar 1 Disorder (BP1): This group consisted of the participants with acute treatment of manic and mixed episodes associated with bipolar 1 disorder who were treated with oral aripiprazole.
- Major Depressive Disorder (MDD): This group consisted of the participants with adjunctive treatment of major depressive disorder who were treated with oral aripiprazole.
- Schizophrenia (SCH): This group consisted of the participants with schizophrenia who were treated with oral aripiprazole.
- Total: Total of all reporting groups
Arm/Group | Bipolar 1 Disorder (BP1) | Major Depressive Disorder (MDD) | Schizophrenia (SCH) | Total
Number analyzed (Participants) | 22 | 12 | 15 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (15.2) | 49.3 (11.2) | 45.5 (11.1) | 46.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 9 | 31
  Male | 7 | 5 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Functionality of an Integrated Call Center for DMS by Adult Subjects With SCH, MDD, or BP1 Who Were Treated With Oral Aripiprazole.
Description: The primary outcome was assessed as the establishment of a functional and operational integrated call center with coordinated feedback to the subject and investigative site to optimize the use of DMS as measured by:
  1. Inbound calls (ie, calls from the subject to the integrated call center) by help type;
  2. Outbound calls (ie, calls from the integrated call center to the subject) by help type.
  The number presented in the table is the number of subjects in trial who made (inbound) or received (outbound) calls
Time Frame: From baseline upto week 9
Population: Intent-to-treat (ITT) Sample: All subjects who entered the trial and used Digital Medicine System (DMS).
Measure: Number; unit: participants
Arm/Group | Bipolar 1 Disorder (BP1) | Major Depressive Disorder (MDD) | Schizophrenia (SCH)
Number analyzed (Participants) | 22 | 12 | 15
participants
  Inbound, Baseline | 0 | 0 | 1
  Inbound, Week 1 | 8 | 8 | 9
  Inbound, Week 2 | 7 | 4 | 6
  Inbound, Week 3 | 2 | 1 | 3
  Inbound, Week 4 | 4 | 2 | 5
  Inbound, Week 5 | 4 | 2 | 4
  Inbound, Week 6 | 0 | 3 | 6
  Inbound, Week 7 | 1 | 3 | 3
  Inbound, Week 8 | 2 | 0 | 4
  Inbound, Week >8 | 0 | 0 | 1
  Outbound, Baseline | 0 | 0 | 0
  Outbound, Week 1 | 22 | 12 | 15
  Outbound, Week 2 | 22 | 12 | 15
  Outbound, Week 3 | 6 | 4 | 3
  Outbound, Week 4 | 6 | 3 | 4
  Outbound, Week 5 | 5 | 3 | 2
  Outbound, Week 6 | 7 | 2 | 5
  Outbound, Week 7 | 9 | 4 | 4
  Outbound, Week 8 | 7 | 5 | 5
  Outbound, Week >8 | 4 | 2 | 0

ADVERSE EVENTS:
Time Frame: 9 Weeks
Arm/Group | Bipolar 1 Disorder (BP1) | Major Depressive Disorder (MDD) | Schizophrenia (SCH)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 10/22 | 9/12 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar 1 Disorder (BP1) (N=22) | Major Depressive Disorder (MDD) (N=12) | Schizophrenia (SCH) (N=15)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.